CLINICAL TRIAL: NCT04703868
Title: A Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of YPI 011 to Rabeprazole in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YJ26-101
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YPI-011 10/500mg (Experimental): Part A: 1 tablet administered before the breakfast during 7 days
  Interventions: Drug: Rabeprazole Sodium 10mg
- YPI-011 20/500mg (Experimental): Part B: 1 tablet administered before the breakfast during 7 days
  Interventions: Drug: Rabeprazole Sodium 20mg

INTERVENTIONS:
Drug: Rabeprazole Sodium 10mg — Part A: 1 tablet administered before the breakfast during 7 days
  Other Names: Reference drug
  Arms: YPI-011 10/500mg
Drug: Rabeprazole Sodium 20mg — Part B: 1 tablet administered before the breakfast during 7 days
  Other Names: Reference drug
  Arms: YPI-011 20/500mg

SUMMARY:
A study to compare the safety, pharmacokinetics and pharmacodynamics of YPI 011 to Rabeprazole in healthy adult subjects

DETAILED DESCRIPTION:
This study is to compare the safety, pharmacokinetics and pharmacodynamics of YPI 011 to Rabeprazole in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Age 19~55 years in healthy volunteers
* BMI is more than 18.0 kg/m^2 , no more than 28.0 kg/m^2
* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who were judged ineligible by the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Integrated gastric acidity | From Day 1 up to Day 28
  Percent decrease from baseline in integrated gastric acidity for 24 hour interval after 7th dose
AUCt,ss | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose

SECONDARY OUTCOMES:
Percent decrease from baseline in integrated gastric acidity for 24 hour interval after 1 st dose | 24 hours
  Evaluateion PD Rabeprazole after multiple dose
Percent of time with gastric pH>4 for 24 hour interval after 1st and 7th dose | From Day 1 up to Day 28
  Evaluateion PD Rabeprazole after multiple dose
Mean and median gastric pH after 1st and 7th dose | From Day 1 up to Day 28
  Evaluateion PD Rabeprazole after multiple dose
AUCτ | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Cmax | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Tmax | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
t1/2 | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
CL/F | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Vz/F | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Cmin,ss, | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Cmax,ss | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Cav,ss, | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Tmax,ss | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
t1/2,ss | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
CLss/F | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Vss/F | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose

CONTACTS AND LOCATIONS:
Overall Officials: Seunghwan Lee, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehak-ro Jongno-gu, South Korea